CLINICAL TRIAL: NCT04583280
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Rilematovir in Infants and Children (≥28 Days to ≤5 Years of Age) and Subsequently in Neonates (<28 Days of Age), Hospitalized With Acute Respiratory Tract Infection Due to Respiratory Syncytial Virus (RSV)
Brief Title: A Study of Rilematovir in Infants and Children and Subsequently in Neonates Hospitalized With Acute Respiratory Tract Infection Due to Respiratory Syncytial Virus (RSV)
Acronym: DAISY
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Janssen made the strategic decision to discontinue the DAISY study. This decision is not based on any safety concerns.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108899; 2020-002023-11 (EudraCT Number); 53718678RSV3001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-10-09; First posted 2020-10-12 (Actual); Results first posted 2023-04-10 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections | interventions — JNJ-53718678

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Rilematovir (Experimental): Participants will receive rilematovir orally based on body weight and age group.
  Interventions: Drug: Rilematovir; Drug: Rilematovir X mg/kg
- Placebo (Experimental): Participants will receive matching placebo of rilematovir based on body weight and age group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rilematovir — Participants of age group greater than or equal to (>=) 28 days to less than (<) 3 months (age group 1) or >= 3 months to < 6 months (age group 2) or >= 6 months to less than or equal to (<=) 5 years (age group 3) will receive rilematovir orally twice a day (BID) from Days 1 to Day 7 or Day 8.
  Other Names: JNJ-53718678
  Arms: Rilematovir
Drug: Rilematovir X mg/kg — Participants of age group birth at term (after at least 37 weeks of gestation) to < 28 days (age group 4) will receive rilematovir orally BID from Days 1 to Day 7 or Day 8. The dose is dependent on outcome of the substudy in neonates and following independent data monitoring (IDMC) review and recommendation.
  Other Names: JNJ-53718678
  Arms: Rilematovir
Drug: Placebo — Participant of age group 1, 2, 3 and 4 will receive matching placebo of rilematovir BID from Days 1 to Day 7 or Day 8 as per assigned age group.
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy of rilematovir compared to placebo treatment with respect to the clinical outcome on the RSV Recovery Scale (RRS).

DETAILED DESCRIPTION:
Respiratory syncytial virus (RSV), a negative-stranded ribonucleic acid (RNA) virus belonging to the Pneumoviridae family, is considered the most important cause of acute lower respiratory tract infection (LRTI) in infants and young children. In most patients, RSV results in upper respiratory tract infection (URTI) eliciting "common cold"-like symptoms, which might last up to 2 weeks, and are usually self-limiting. RSV-related LRTI is a major cause of hospital admissions and death in young children worldwide. Rilematovir is an investigational, small molecule, RSV fusion inhibitor. This study aims to evaluate the efficacy and safety of rilematovir in hospitalized infants and children (greater than or equal to [>=] 28 days to less than or equal to [<=] 5 years) and, subsequent to completion of the neonatal substudy, in hospitalized neonates (born at term, less than [<] 28 days of age) with RSV infection. The study will include a Screening Period, a Treatment Period, and a Follow-up Period. The total study duration for each participant will be approximately 36 days (Screening included). The efficacy assessments include evaluation under the RRS and the safety assessments include evaluations of physical examinations, vital signs, electrocardiograms, clinical laboratory tests, and adverse events.

ELIGIBILITY:
Inclusion criteria:

* The participant weighs within greater than or equal to (>=) 2.4 kilograms (kg) and less than or equal to (<=) 24.6 kg
* Each participant's parent(s) (preferably both if available or as per local requirements) or their legally acceptable representative(s) has/have signed an informed consent form (ICF) indicating that (s)he understands the purpose of, and procedures required for, the study; is willing for their child to participate in the study; with regards to the concomitant medication, the lifestyle consideration and study procedures and assessments to be performed by the parent(s)/caregiver(s) as well as those by the investigator/study site personnel
* The participant has an acute respiratory illness with at least 1 of the signs/symptoms within 24 hours prior to start of screening and at screening, as evaluated by the investigator in Upper respiratory tract infection: nasal congestion or rhinorrhea; and Lower respiratory tract infection: increased respiratory effort (as evidenced by subcostal, intercostal or tracheosternal retractions, grunting, head bobbing, nasal flaring, or tachypnea), wheezing, cough, cyanosis, or apnea; and systemic/general: feeding difficulties (defined as <75 percent [%] intake of normal food amounts); dehydration; fever; disturbed sleep, or disturbed activity level (irritable/restless/agitated/less responsive). Cough or wheezing cannot be the only LRTI sign/symptom present, that is, at least one other LRTI sign/symptom needs to be present for eligibility
* The time of onset of RSV signs/symptoms to the anticipated time of randomization must be less than or equal to (<=) 3 days. Onset of signs/symptoms is defined as the time of the day (or part of the day if time of the day cannot be specified) the parent(s)/caregiver(s) became aware of the first sign and/or symptom consistent with respiratory or systemic/general manifestation of signs/symptoms of RSV infection. The time of sign/symptom onset has to be assessed as accurately as possible
* Participants are otherwise healthy or have (a) risk factor(s) for severe RSV disease

Exclusion criteria:

* The participant has had either confirmed severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) infection (test positive) during the four weeks prior to randomization, or close contact with a person with COVID-19 (test confirmed or suspected SARS CoV-2 infection) within 14 days prior to randomization
* Confirmed QT interval corrected for heart rate according to Fridericia's formula (QTcF) interval greater than (>) 450 milliseconds (msec) per the machine read parameter result at screening. Presence of an abnormal QTcF interval should be confirmed by repeat electrocardiogram (ECG) recording during screening
* Known personal or family history of Long QT Syndrome or sudden cardiac death
* Presence of repetitive ventricular premature contractions (>10/minutes [min]), second- or third-degree heart block, or complete or incomplete left bundle branch block, or complete right bundle branch block per the machine read ECG result at screening. Presence of any of the above abnormalities should be confirmed by repeat ECG recording during screening

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (142):
- United States (5):
  - Arnold Palmer Hospital For Children, Orlando, Florida
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Jacobi Medical Center, The Bronx, New York
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - MultiCare Health Systems for Research and Innovation, Tacoma, Washington
- Argentina (7):
  - Hospital Interzonal General de Agudos Dr. Jose Penna, Bahía Blanca
  - Hospital Italiano Regional Del Sur, Bahía Blanca
  - Hospital General de Niños Pedro de Elizalde, Buenos Aires
  - Hospital Universitario Austral, Pilar
  - Instituto Medico Rio Cuarto, Río Cuarto
  - Hospital del Niño Jesús, San Miguel de Tucumán
  - Clinica Mayo de UMCB, San Miguel de Tucumán
- Belgium (5):
  - ULB Hôpital Erasme, Anderlecht
  - AZ Sint Jan Brugge Oostende AV, Bruges
  - UZ Brussel, Brussels
  - Cliniques Universitaires Saint Luc, Brussels
  - UZ Leuven, Leuven
- Brazil (9):
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte
  - Fundacao para o Desenvolvimento Medico Hospitalar (UNESP Botucatu), Botucatu
  - Sociedade Campineira de Educacao e Instrucao Hospital e Maternidade Celso Pierro, Campinas
  - Nucleo de Pesquisa do Hospital Pequeno Princípe, Curitiba
  - Secretaria da Saude do Estado do Ceara - Hospital Doutor Carlos Alberto Studart Gomes, Fortaleza
  - Associacao Hospitalar Moinhos de Vento, Porto Alegre
  - Hospital Das Clinicas Da Faculdade De Medicina De RPUSP HCRP, Ribeirão Preto
  - Fundacao Jose Luiz Egydio Setubal, São Paulo
  - Santa Casa de Misericórdia de Votuporanga, Votuporanga
- Bulgaria (5):
  - UMHAT 'Sveti Georgi'-Plovdiv, Plovdiv
  - UMHAT 'Kanev' EAD, Rousse
  - Acibadem City Clinic Tokuda Hospital, Sofia
  - UMHAT 'Aleksandrovska' EAD, Sofia
  - SHATCD 'Prof. Ivan Mitev' EAD, Sofia
- China (5):
  - Capital Institute of Pediatrics, Beijing
  - Beijing Children's Hospital, Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - West China Second University Hospital, Sichuan University, Chengdu
  - Guangzhou Women And Children's Medical Center, Guangzhou
- Czechia (3):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Thomayerova nemocnice, Prague
- Estonia (2):
  - Tallinn Children's Hospital, Tallinn
  - Tartu University Hospital, Tartu
- Germany (3):
  - Universitätsklinik Freiburg, Freiburg im Breisgau
  - HELIOS Klinikum Wuppertal GmbH, Wuppertal
  - Universitatsklinikum Wurzburg, Würzburg
- Hungary (8):
  - Semmelweis Egyetem, II. sz. Gyermekgyógyászati Klinika, Budapest
  - Bethesda Gyermekkórház, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Bacs-kiskun Megyei Korhaz, Kecskemét
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi Oktato Korhaz, Miskolc
  - Szegedi Tudomanyegyetem, Szeged
  - Csolnoky Ferenc Korhaz, Veszprém
- Israel (5):
  - Soroka University Medical Center, Beersheba
  - Ruth Rappaport Children's Hospital, Rambam Health Care Campus, Haifa
  - Schneider Children's Medical Center, Petah Tikva
  - Pediatrics B, Safra Children's Hospital, Tel Hashomer, Ramat Gan
  - Sourasky MC, Tel Aviv
- Italy (4):
  - A O U Sant Orsola Malpighi, Bologna
  - Università degli Studi di Milano, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Department of Pediatrics University of Pavia, Policlinico San Matteo, Pavia
  - Ospedale degli Infermi, Ponderano
- Japan (15):
  - Fukui Prefectural Hospital, Fukui-shi
  - Fukuyama City Hospital, Fukuyama
  - Kagoshima Children's Hospital, Hioki
  - Teine Keijinkai Hospital, Hokkaido
  - National Hospital Organization Kanazawa Medical Center, Ishikawa
  - Japan Community Health care Organization Kyushu Hospital, Kitakyushu-shi
  - Kobe City Medical Center General Hospital, Kobe
  - Kochi Health Sciences Center, Kochi
  - Maebashi Red Cross Hospital, Maebashi
  - Kojunkai Daido Hospital, Nagoya
  - National Hospital Organization Niigata National Hospital, Niigata
  - National Hospital Organization Beppu Medical Center, Ōita
  - National Hospital Organization Saitama National Hospital, Saitama
  - National Hospital Organization Ureshino Medical Center, Ureshino-shi
  - Yamanashi Prefectural Central Hospital, Yamanashi
- Children's Clinical University Hospital, Riga, Latvia
- Malaysia (5):
  - Hospital Selayang, Batu Caves
  - Hospital Bintulu, Bintulu
  - Hospital Miri, Miri
  - Hospital Sibu, Sibu
  - Hospital Taiping, Taiping
- Mexico (4):
  - Instituto Nacional de Pediatría, Mexico City
  - Hospital Infantil de Mexico Federico Gomez, Mexico City
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey
  - Centro Medico Zambrano Hellion, Monterrey
- Cevaxin Avenida Mexico, Panama City, Panama
- Poland (4):
  - Krakowski Szpital Specjalistyczny im Jana Pawla II, Krakow
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im M Kopernika w Lodzi, Lodz
  - Uniwersytecki Szpital Dzieciecy w Lublinie, Lublin
  - Dzieciecy Szpital Kliniczny im Jozefa Polikarpa Brudzinskiego, Warsaw
- Slovakia (2):
  - DFNsP Banska Bystrica, Banská Bystrica
  - Pediatric Pulmonology Clinic, University Hospital Bratislava, Bratislava
- South Korea (7):
  - Kyungpook National University Hospital, Daegu
  - CHA Bundang Medical Center, CHA University, Gyeonggi-do
  - Korea Institute of Radiological and Medical Sciences, Seoul
  - Nowon Eulji Medical Center, Eulji University, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Inje University Sanggye Paik Hospital, Seoul
- Spain (14):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp. Univ. de Cruces, Barakaldo
  - Hosp Reina Sofia, Córdoba
  - Hosp. Univ. de Getafe, Getafe
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp. Univ. Hm Monteprincipe, Madrid
  - Hosp. Univ. Severo Ochoa, Madrid
  - Hosp. Univ. Pta. de Hierro Majadahonda, Majadahonda
  - Hosp. Puerta Del Sur, Móstoles
  - Complejo Hosp. de Navarra, Pamplona
  - Hosp. Quiron Madrid Pozuelo, Pozuelo de Alarcón
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela
- Astrid Lindgrens barnsjukhus Solna, Stockholm, Sweden
- Taiwan (5):
  - Hsinchu MacKay Memorial Hospital, Hsinchu
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Chang Gung Medical Foundation, Taoyuan
- Thailand (6):
  - Tropical Medicine Hospital, Mahidol University, Bangkok
  - Siriraj Hospital Mahidol University, Bangkok
  - Maharaj Nakorn Chiangmai Hospital, Chiang Mai
  - Srinagarind Hospital, Khon Kaen
  - Bamrasnaradura Infectious Disease Institute, Nonthaburi
  - Faculty of Medicine Chulalongkorn University, Pathumwan
- Turkey (Türkiye) (7):
  - Cukurova University Medical Faculty Balcali Hospital, Adana
  - Hacettepe University Medical Faculty, Ankara
  - Gazi University Medical Faculty, Ankara
  - Istanbul University Istanbul Medical Faculty, Istanbul
  - Ege University Medical Faculty, Izmir
  - Saglik Bilimleri University Sariyer Hamidiye Etfal Training and Research Hospital, Sarıyer
  - Karadeniz Teknik University Medical Faculty, Trabzon
- Ukraine (9):
  - MNPE City Children's Clinical Hospital № 6 of Dnipro City Council, Dnipro
  - ME 'Dnipropetrovsk Regional Children's Clinical Hospital of Dnipropetrovsk Regional Council', Dnipro
  - Kharkiv National Medical University on based CHPI Kharkiv Municipal Clinical Children's Hospital 16, Kharkiv
  - MUNICIPAL NON-PROFIT ENTERPRISE 'Kryvyi Rih CITY HOSPITAL №16' Kryvyi Rih CITY COUNCIL, Kryvyi Rih
  - Odessa Regional Child Hospital, Odesa
  - SSU Division MU Ch of pediatrics of PGE with propedeutic pediatrics and children infections course, Sumy
  - Sumy Regional Childrens Clinical Hospital, Sumy
  - Municipal institution 'Vinnytsia Regional Clinical Children's Infectious Diseases Hospital', Vinnytsia
  - MNPE Zaporizhzhya Regional Clinical Children's Hospital of Zaporizhzhya Regional Council, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 28 participants with acute respiratory tract infection due to respiratory syncytial virus (RSV) were randomized and treated (8 participants in placebo arm and 20 participants in rilematovir arm). Of these, 27 participants completed the study.
Groups:
- Placebo: Participants aged greater than or equal to (>=) 28 days to less than (<) 3 months, >=3 to <6 months, and >=6 months to less than or equal to (<=) 5 years received placebo matching to rilematovir as oral suspension twice daily (BID) from Days 1 to 7 (14 consecutive doses).
- Rilematovir: Participants aged >=28 days to <3 months, >=3 to <6 months, and >=6 months to <=5 years received rilematovir 2.5 milligrams per kilogram (mg/kg), 3 mg/kg and 4.5 mg/kg respectively, as oral suspension BID from Days 1 to 7 (14 consecutive doses).
Period: Overall Study
Arm/Group | Placebo | Rilematovir
Started | 8 | 20
Completed | 8 | 19
Not Completed | 0 | 1
Not completed — Consent withdrawn by parent/caregiver | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rilematovir | Total
Number analyzed (Participants) | 8 | 20 | 28
Age, Continuous [Mean (Standard Deviation); unit: months] | 15.3 (19.4) | 16.2 (13.67) | 15.9 (15.14)
Age, Customized [Count of Participants; unit: Participants]
  Infants and toddlers(28 days-23 months) | 6 | 14 | 20
  Children (2-11 years) | 2 | 6 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 12 | 18
  Male | 2 | 8 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 8 | 11
  Not Hispanic or Latino | 5 | 8 | 13
  Unknown or Not Reported | 0 | 4 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 1 | 3
  Black or African American | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 6 | 14 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
  Missing | 0 | 1 | 1
  Other | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants by Respiratory Syncytial Virus (RSV) Recovery Scale (RRS) Category
Description: RRS was an ordinal scale to assess a participant's clinical status. The RRS provided 7 mutually exclusive categories ordered from best (1) to worst (7) where 1 =home without signs/symptoms, 2 =home with sign/symptoms, 3 =ward without supplemental oxygen (O2) or feeding/hydration, 4 =ward with supplemental or feeding/hydration, 5 =intensive care unit (ICU) without mechanical ventilation (included both invasive and non-invasive mechanical ventilation), 6 =required mechanical ventilation and 7=worst (death). Higher category indicates worse condition. With or without signs/symptoms was defined as the key RSV signs/symptoms (breathing problems, retractions, tachypnea, cough, wheezing/breathing sounds, and tachycardia) resolved (absent or mild) or not resolved assessed by parent/caregiver.
Time Frame: Baseline to Day 8
Population: Intent to treat - infected (ITT-i) analysis set included all randomized participants who received at least 1 dose of study intervention and had an RSV infection confirmed by central laboratory analysis. Due to the early termination of study, last day of RRS treatment (Day 8) was considered instead of the original planned day defined as when 50% participants would have been discharged.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rilematovir
Number analyzed (Participants) | 8 | 19
Percentage of participants
  Home without symptoms | 25.0 | 31.6
  Home with symptoms | 50.0 | 26.3
  Ward without supplemental oxygen/feeding/hydration | 25.0 | 36.8
  Ward with supplemental or feeding/hydration | 0 | 5.3
  ICU without mechanical ventilation | 0 | 0
  Requiring mechanical ventilation | 0 | 0
  Death | 0 | 0

2. Secondary Outcome: Percentage of Participants Clinically Resolved From RSV Disease Based on the Clinician Reported Outcome (ClinRO) Sign/Symptoms at Day 8
Description: Clinically resolved was defined as participant required no oxygen supplementation, no supplemental feeding/hydration, no need for ICU and had Key RSV signs/symptoms resolved to absent or mild as per ClinRO signs/symptoms. Clinically resolved Key RSV signs/symptoms were assessed based on clinician's observations as resolved if participant had no retractions, tachypnea, tachycardia, breathing problems (nasal flaring, head bobbing, grunting); cough (resolved if little or no coughing or occasional strong cough or sometimes productive) and wheezing (resolved if no wheezing or terminal expiratory wheezing or only with stethoscope).
Time Frame: Day 8
Population: ITT-i analysis set included all randomized participants who received at least 1 dose of study intervention and had an RSV infection confirmed by central laboratory analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rilematovir
Number analyzed (Participants) | 8 | 19
Percentage of participants | 37.5 | 31.6

3. Secondary Outcome: Time From First Study Dose to Resolution of Key RSV Signs/Symptoms Based on Observer Reported Outcome (ObsRO) After Free of Supplementation (Oxygen/Feeding/Hydration) for at Least 24 Hours
Description: Time (in hours) from first dose of study intervention to first resolution of key RSV signs/symptoms was evaluated based on ObsRO assessment after free of supplementation (O2/feeding/hydration) for at least 24 hours. Clinically resolved was defined as participant required no oxygen supplementation, no supplemental feeding/hydration, no need for ICU and had key RSV signs/symptoms resolved to absent or mild as per ObsRO signs/symptoms. Resolution of key signs/symptoms assessment was based on observations of child's parent/caregiver as resolved if no retractions, tachypnea, tachycardia, breathing problems (gasping for air nostrils, flaring when breathing, head bobbed back and forth when breathing), no breathing sound; cough (no coughing, little coughing without problems). Kaplan-Meier method was used for estimation.
Time Frame: Up to Day 21
Population: ITT-i analysis set included all randomized participants who received at least 1 dose of study intervention and had RSV infection confirmed by central laboratory analysis.
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Placebo | Rilematovir
Number analyzed (Participants) | 8 | 19
Hours | 237.0 [114.38 to NA] — Here, NA indicates that upper limit of 95% confidence interval (CI) could not be estimated due to low number of participants with events. | 144.8 [96.09 to 210.93]

4. Secondary Outcome: Number of Participants With Post-baseline RSV-related Complications
Description: RSV related complications included respiratory complications (respiratory failure, apnoeic attacks, bronchiolitis, bronchial obstruction, pneumonia and asthmatic crisis), infectious complications (otitis media, bacterial respiratory tract infections and sepsis), cardiovascular complications (arrhythmia, cardiogenic shock, hemodynamic instability, congestive cardiac failure), acid-base or electrolyte complications (metabolic acidosis, metabolic alkalosis, hyponatremia, hypokalemia, hyperkalemia, hypocalcemia, hypercalcemia, hypoglycemia and hyperglycemia). Participants were counted only once, regardless of the number of complications they actually experienced.
Time Frame: Up to Day 35
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rilematovir
Number analyzed (Participants) | 8 | 19
Participants | 1 | 3

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product and did not necessarily have a causal relationship with the treatment. A TEAE was defined as an AE with an onset after the initiation study drug (Day 1) up to end of study (Day 35). AEs included both serious and non-serious AEs.
Time Frame: Day 1 up to Day 35
Population: Safety analysis set included all participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rilematovir
Number analyzed (Participants) | 8 | 20
Participants | 5 | 11

6. Secondary Outcome: Number of Participants With Abnormalities in Clinical Laboratory Values
Description: Number of participants with abnormally low (AL) and abnormally high (AH) values of bicarbonate, direct bilirubin, urea nitrogen, basophils, eosinophils, erythrocyte (Ery). mean corpuscular hemoglobin (HGB) concentration (conc), Ery. mean corpuscular hemoglobin, erythrocytes, leukocytes, lymphocytes, monocytes, neutrophils and reticulocytes were reported based on the investigator's discretion.
Time Frame: Up to Day 35
Population: Safety analysis set included all participants who received at least 1 dose of study intervention. Here, N (Overall number of participants analyzed) signifies participants evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants with available data at each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rilematovir
Number analyzed (Participants) | 8 | 18
Participants
  Bicarbonate- Abnormally low: number analyzed (Participants) | 8 | 17
  Bicarbonate- Abnormally low | 1 | 3
  Bicarbonate- Abnormally high: number analyzed (Participants) | 8 | 17
  Bicarbonate- Abnormally high | 0 | 0
  Direct bilirubin- Abnormally low: number analyzed (Participants) | 7 | 16
  Direct bilirubin- Abnormally low | 2 | 9
  Direct bilirubin- Abnormally high: number analyzed (Participants) | 7 | 16
  Direct bilirubin- Abnormally high | 0 | 0
  Urea nitrogen- Abnormally low: number analyzed (Participants) | 8 | 17
  Urea nitrogen- Abnormally low | 1 | 3
  Urea nitrogen- Abnormally high: number analyzed (Participants) | 8 | 17
  Urea nitrogen- Abnormally high | 0 | 0
  Basophils- Abnormally low: number analyzed (Participants) | 7 | 17
  Basophils- Abnormally low | 0 | 0
  Basophils- Abnormally high: number analyzed (Participants) | 7 | 17
  Basophils- Abnormally high | 0 | 1
  Eosinophils- Abnormally low: number analyzed (Participants) | 7 | 17
  Eosinophils- Abnormally low | 0 | 0
  Eosinophils- Abnormally high: number analyzed (Participants) | 7 | 17
  Eosinophils- Abnormally high | 5 | 12
  Ery. mean corpuscular HGB conc.-AL: number analyzed (Participants) | 7 | 17
  Ery. mean corpuscular HGB conc.-AL | 1 | 3
  Ery. mean corpuscular HGB conc.-AH: number analyzed (Participants) | 7 | 17
  Ery. mean corpuscular HGB conc.-AH | 0 | 0
  Ery. mean corpuscular hemoglobin-AL: number analyzed (Participants) | 7 | 18
  Ery. mean corpuscular hemoglobin-AL | 0 | 3
  Ery. mean corpuscular hemoglobin-AH: number analyzed (Participants) | 7 | 18
  Ery. mean corpuscular hemoglobin-AH | 0 | 0
  Erythrocytes- Abnormally low: number analyzed (Participants) | 7 | 18
  Erythrocytes- Abnormally low | 0 | 0
  Erythrocytes- Abnormally high: number analyzed (Participants) | 7 | 18
  Erythrocytes- Abnormally high | 0 | 2
  Leukocytes- Abnormally low: number analyzed (Participants) | 7 | 18
  Leukocytes- Abnormally low | 1 | 1
  Leukocytes- Abnormally high: number analyzed (Participants) | 7 | 18
  Leukocytes- Abnormally high | 0 | 5
  Lymphocytes- Abnormally low: number analyzed (Participants) | 7 | 17
  Lymphocytes- Abnormally low | 0 | 0
  Lymphocytes- Abnormally high: number analyzed (Participants) | 7 | 17
  Lymphocytes- Abnormally high | 0 | 3
  Monocytes- Abnormally low: number analyzed (Participants) | 7 | 17
  Monocytes- Abnormally low | 1 | 4
  Monocytes- Abnormally high: number analyzed (Participants) | 7 | 17
  Monocytes- Abnormally high | 0 | 0
  Neutrophils- Abnormally low: number analyzed (Participants) | 7 | 17
  Neutrophils- Abnormally low | 4 | 10
  Neutrophils- Abnormally high: number analyzed (Participants) | 7 | 17
  Neutrophils- Abnormally high | 0 | 0
  Reticulocytes- Abnormally low: number analyzed (Participants) | 7 | 18
  Reticulocytes- Abnormally low | 0 | 0
  Reticulocytes- Abnormally high: number analyzed (Participants) | 7 | 18
  Reticulocytes- Abnormally high | 1 | 1

7. Secondary Outcome: Number of Participants With Abnormalities in Electrocardiograms (ECGs)
Description: Number of participants with abnormally low and abnormally high values of ECG parameters (PR interval and RR interval) as assessed based on the investigator's discretion were reported.
Time Frame: Up to Day 35
Population: Safety analysis set included all participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rilematovir
Number analyzed (Participants) | 8 | 20
Participants
  PR Interval- Abnormally low | 0 | 0
  PR Interval- Abnormally high | 0 | 1
  RR Interval- Abnormally low | 1 | 7
  RR Interval- Abnormally high | 0 | 0

8. Secondary Outcome: Number of Participants With Abnormalities in Vital Signs
Description: Number of participants with abnormally low and abnormally high values of vital signs from baseline were assessed based on investigator's discretion. Vital signs included systolic blood pressure (SBP) (millimeter of mercury [mmHg]), diastolic blood pressure (DBP) (mmHg), pulse rate (beats per minute), respiratory rate (breaths per minute), temperature (degree Celsius) and oxygen saturation (in percentage).
Time Frame: Up to Day 35
Population: Safety analysis set included all participants who received at least 1 dose of study intervention. Here, 'n' (number analyzed) signifies number of participants with available data at each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rilematovir
Number analyzed (Participants) | 8 | 20
Participants
  SBP- Abnormally low | 0 | 0
  SBP- Abnormally high | 0 | 4
  DBP- Abnormally low | 0 | 0
  DBP- Abnormally high | 1 | 3
  Pulse Rate- Abnormally low | 0 | 0
  Pulse Rate- Abnormally high | 1 | 2
  Respiratory Rate- Abnormally low | 0 | 0
  Respiratory Rate- Abnormally high | 0 | 3
  Temperature - Abnormally low | 0 | 0
  Temperature - Abnormally high | 1 | 0
  Oxygen Saturation- Abnormally low: number analyzed (Participants) | 8 | 19
  Oxygen Saturation- Abnormally low | 0 | 1
  Oxygen Saturation- Abnormally high: number analyzed (Participants) | 8 | 19
  Oxygen Saturation- Abnormally high | 0 | 0

9. Secondary Outcome: Percentage of Participants Requiring Intensive Care Unit (ICU) Stay After First Dose of Rilematovir
Description: Percentage of participants requiring ICU stay was analyzed and reported.
Time Frame: Up to Day 35
Population: ITT-i analysis set included all randomized participants who received at least 1 dose of study intervention and had an RSV infection confirmed by central laboratory analysis. Here, N (Overall number of participants analyzed) signifies participants with no ICU stay before first dose of rilematovir.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Rilematovir
Number analyzed (Participants) | 6 | 17
Percentage of Participants | 0 | 0

10. Secondary Outcome: Duration of ICU Stay
Description: Duration (in hours) of ICU stay was defined as total number of hours a participant experienced an ICU stay from first dose of rilematovir until study termination, calculated as the sum of all separate records of ICU stay.
Time Frame: Up to Day 35
Population: ITT-i analysis set included all randomized participants who received at least 1 dose of study intervention and had an RSV infection confirmed by central laboratory analysis. Here, N (Overall number of participants analyzed) signifies participants who required ICU stay before first dose of rilematovir and continued after first dose plus participants who required ICU stay after first dose of drug without prior ICU stay.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | Rilematovir
Number analyzed (Participants) | 2 | 2
hours | 66.46 (24.145) [lower limit 24.145] | 40.83 (22.822) [lower limit 22.822]

11. Secondary Outcome: Percentage of Participants Requiring Re-hospitalization for Respiratory/Other Reasons
Description: Percentage of participants requiring re-hospitalization (participants re-hospitalized [ward or ICU] after been discharged from hospital) for respiratory/other reasons were reported.
Time Frame: Up to Day 35
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rilematovir
Number analyzed (Participants) | 8 | 19
Percentage of participants | 0 | 0

12. Secondary Outcome: Percentage of Participants Requiring Oxygen Supplementation After First Dose of Rilematovir
Description: Percentage of participants requiring any type of oxygen supplementation (invasive mechanical ventilation, non-invasive mechanical ventilation and non-invasive non-mechanical ventilation) were reported.
Time Frame: Up to Day 35
Population: ITT-i analysis set included all randomized participants who received at least 1 dose of study intervention and had an RSV infection confirmed by central laboratory analysis. Here, N (overall number of participants analyzed) signifies participants with no use of oxygen supplementation before first dose of rilematovir.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rilematovir
Number analyzed (Participants) | 6 | 13
Percentage of participants | 16.7 | 30.8

13. Secondary Outcome: Duration of Oxygen Supplementation
Description: Duration (in hours) of oxygen supplementation was defined as total number of hours a participant used supplemental oxygen from either prior to first dose and/or after first dose of drug until study termination, calculated as the sum of all separate records of supplementation.
Time Frame: Up to Day 35
Population: ITT-i analysis set included all randomized participants who received at least 1 dose of study intervention and had an RSV infection confirmed by central laboratory analysis. Here, N (Overall number of participants analyzed) signifies participants who required oxygen supplementation before first dose of rilematovir and continued after first dose plus participants who required oxygen supplementation after first dose of rilematovir without prior oxygen supplementation.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Placebo | Rilematovir
Number analyzed (Participants) | 3 | 10
Hours | 39.91 (26.146) [lower limit 26.146] | 66.59 (51.956) [lower limit 51.956]

14. Secondary Outcome: Percentage of Participants Requiring Hydration and/or Feeding by Intravenous (IV) Administration or Nasogastric Tube After First Dose of Rilematovir
Description: Percentage of participants requiring any type of hydration and/or feeding by intravenous (IV) administration or nasogastric tube or percutaneous endoscopic gastrostomy was reported.
Time Frame: Up to Day 35
Population: ITT-i analysis set included all randomized participants who received at least 1 dose of study intervention and had an RSV infection confirmed by central laboratory analysis. Here, N (Overall number of participants analyzed) signifies participants with no use of feeding/hydration supplementation before 1st dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rilematovir
Number analyzed (Participants) | 3 | 15
Percentage of participants | 33.3 | 0

15. Secondary Outcome: Duration of Supplemental Feeding/Hydration
Description: Duration (in hours) of supplemental feeding/hydration was defined as total number of hours a participant was administered feeding/hydration supplementation from either prior to first dose and/or after first dose of drug until study termination, calculated as the sum all separate records of supplementation use per participant.
Time Frame: Up to Day 35
Population: ITT-i analysis set included all randomized participants who received at least 1 dose of study intervention and had an RSV infection confirmed by central laboratory analysis. Here, N (Overall number of participants analyzed) signifies participants who required supplemental feeding/hydration before first dose of rilematovir and continued after first dose plus participants who required supplemental feeding/hydration after first dose of rilematovir without prior supplemental feeding/hydration.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Placebo | Rilematovir
Number analyzed (Participants) | 6 | 4
Hours | 43.13 (41.526) | 31.96 (21.311)

16. Secondary Outcome: Number of Participants With Medical Encounters and Treatments
Description: Medical resource utilization was assessed by medical care encounters and treatments. Medical encounters and treatments included physician or emergency room visits, tests and procedures, and medications, surgeries and other selected procedures, inpatient and outpatient.
Time Frame: Up to Day 35
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rilematovir
Number analyzed (Participants) | 8 | 19
Participants | 1 | 3

17. Secondary Outcome: RSV Viral Load at Baseline, Days 2, 3, 5, 8, 14 and 21
Description: Antiviral activity was determined based on measurements of RSV viral load which was measured by quantitative reverse transcription polymerase chain reaction (qRT-PCR) in the mid-turbinate (MT) nasal swab specimens.
Time Frame: Baseline, Days 2, 3, 5, 8, 14 and 21
Population: ITT-i analysis set included all randomized participants who received at least 1 dose of study intervention and had an RSV infection confirmed by central laboratory analysis. Here, 'n' (number analyzed) signifies number of participants with data evaluable at each specified time point.
Measure: Mean (Standard Deviation); unit: log10 copies per milliliter
Arm/Group | Placebo | Rilematovir
Number analyzed (Participants) | 8 | 19
log10 copies per milliliter
  Baseline: number analyzed (Participants) | 8 | 18
  Baseline | 7.031 (1.9995) | 6.286 (1.3671)
  Day 2 | 6.000 (1.5678) | 5.579 (1.5668)
  Day 3 | 5.465 (1.7454) | 4.981 (1.9530)
  Day 5 | 4.066 (1.5565) | 4.132 (1.5199)
  Day 8: number analyzed (Participants) | 8 | 18
  Day 8 | 1.373 (2.0865) | 2.156 (2.1681)
  Day 14: number analyzed (Participants) | 7 | 17
  Day 14 | 1.217 (2.1478) | 0.709 (1.3389)
  Day 21: number analyzed (Participants) | 7 | 17
  Day 21 | 0.414 (1.0961) | 0.464 (1.4547)

18. Secondary Outcome: Change From Baseline in RSV Viral Load at Days 2, 3, 5, 8, 14 and 21
Description: Antiviral activity was determined based on measurements of RSV viral load which was measured by qRT-PCR in the MT nasal swab specimens.
Time Frame: Baseline, Days 2, 3, 5, 8, 14 and 21
Population: ITT-i analysis set included all randomized participants who received at least 1 dose of study intervention and had an RSV infection confirmed by central laboratory analysis. Here, N (Overall number of participants analyzed) signifies participants evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants with data evaluable at each specified time point.
Measure: Mean (Standard Deviation); unit: log10 copies per milliter
Arm/Group | Placebo | Rilematovir
Number analyzed (Participants) | 8 | 18
log10 copies per milliter
  Day 2 | -1.031 (0.6091) | -0.825 (1.2906)
  Day 3 | -1.566 (2.2167) | -1.436 (1.5185)
  Day 5 | -2.965 (1.9154) | -2.241 (1.3393)
  Day 8: number analyzed (Participants) | 8 | 17
  Day 8 | -5.658 (1.9872) | -4.126 (1.8461)
  Day 14: number analyzed (Participants) | 7 | 17
  Day 14 | -5.693 (2.2654) | -5.640 (2.0261)
  Day 21: number analyzed (Participants) | 7 | 16
  Day 21 | -7.207 (1.3201) | -5.789 (1.9560)

19. Secondary Outcome: Percentage of Participants With Undetectable RSV Viral Load
Description: Percentage of participants with undetectable RSV viral load was analyzed.
Time Frame: Baseline, Days 2, 3, 5, 8, 14 and 21
Population: as for outcome 17
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Rilematovir
Number analyzed (Participants) | 8 | 19
Percentage of Participants
  Baseline: number analyzed (Participants) | 8 | 18
  Baseline | 0 | 0
  Day 2 | 0 | 0
  Day 3 | 0 | 5.3
  Day 5 | 0 | 0
  Day 8: number analyzed (Participants) | 8 | 18
  Day 8 | 62.5 | 44.4
  Day 14: number analyzed (Participants) | 7 | 17
  Day 14 | 71.4 | 76.5
  Day 21: number analyzed (Participants) | 7 | 17
  Day 21 | 85.7 | 88.2

20. Secondary Outcome: Plasma Concentrations of Rilematovir
Description: Plasma concentrations of rilematovir were assessed. Participant wise data were reported for this outcome measure.
Time Frame: 1 hour Post-dose (Day 1) and pre-dose (Day 2)
Population: Pharmacokinetics analysis set (PKAS) included participants who had received at least 1 dose of rilematovir and had at least 1 valid blood sample drawn for pharmacokinetics analysis. No summary analysis was done as study was terminated early and participant wise data were reported. Here, "n" (Number analyzed) signifies specific participant with data evaluable at each specified timepoint.
Measure: Number; unit: nanogram per milliliter
Arm/Group | Rilematovir
Number analyzed (Participants) | 18
nanogram per milliliter
  Participant 1 Day 1: number analyzed (Participants) | 1
  Participant 1 Day 1 | 1450
  Participant 2 Day 1: number analyzed (Participants) | 1
  Participant 2 Day 1 | 1750
  Participant 3 Day 1: number analyzed (Participants) | 1
  Participant 3 Day 1 | 72.5
  Participant 4 Day 1: number analyzed (Participants) | 1
  Participant 4 Day 1 | 656
  Participant 5 Day 1: number analyzed (Participants) | 1
  Participant 5 Day 1 | 918
  Participant 6 Day 1: number analyzed (Participants) | 1
  Participant 6 Day 1 | 1050
  Participant 7 Day 1: number analyzed (Participants) | 1
  Participant 7 Day 1 | 135
  Participant 8 Day 1: number analyzed (Participants) | 1
  Participant 8 Day 1 | 1730
  Participant 9 Day 1: number analyzed (Participants) | 1
  Participant 9 Day 1 | 602
  Participant 10 Day 1: number analyzed (Participants) | 1
  Participant 10 Day 1 | 1810
  Participant 11 Day 1: number analyzed (Participants) | 1
  Participant 11 Day 1 | 1640
  Participant 12 Day 1: number analyzed (Participants) | 1
  Participant 12 Day 1 | 3760
  Participant 13 Day 1: number analyzed (Participants) | 1
  Participant 13 Day 1 | 561
  Participant 14 Day 1: number analyzed (Participants) | 1
  Participant 14 Day 1 | 127
  Participant 15 Day 1: number analyzed (Participants) | 1
  Participant 15 Day 1 | 787
  Participant 16 Day 1: number analyzed (Participants) | 1
  Participant 16 Day 1 | 2020
  Participant 17 Day 1: number analyzed (Participants) | 1
  Participant 17 Day 1 | 157
  Participant 18 Day 1: number analyzed (Participants) | 1
  Participant 18 Day 1 | 1260
  Participant 1 Day 2: number analyzed (Participants) | 1
  Participant 1 Day 2 | 134
  Participant 2 Day 2: number analyzed (Participants) | 1
  Participant 2 Day 2 | 281
  Participant 3 Day 2: number analyzed (Participants) | 1
  Participant 3 Day 2 | 5.74
  Participant 5 Day 2: number analyzed (Participants) | 1
  Participant 5 Day 2 | 417
  Participant 6 Day 2: number analyzed (Participants) | 1
  Participant 6 Day 2 | 828
  Participant 7 Day 2: number analyzed (Participants) | 1
  Participant 7 Day 2 | 1030
  Participant 8 Day 2: number analyzed (Participants) | 1
  Participant 8 Day 2 | 339
  Participant 9 Day 2: number analyzed (Participants) | 1
  Participant 9 Day 2 | 186
  Participant 10 Day 2: number analyzed (Participants) | 1
  Participant 10 Day 2 | 687
  Participant 11 Day 2: number analyzed (Participants) | 1
  Participant 11 Day 2 | 1750
  Participant 12 Day 2: number analyzed (Participants) | 1
  Participant 12 Day 2 | 4650
  Participant 13 Day 2: number analyzed (Participants) | 1
  Participant 13 Day 2 | 311
  Participant 14 Day 2: number analyzed (Participants) | 1
  Participant 14 Day 2 | 77.3
  Participant 15 Day 2: number analyzed (Participants) | 1
  Participant 15 Day 2 | 749
  Participant 16 Day 2: number analyzed (Participants) | 1
  Participant 16 Day 2 | 457
  Participant 17 Day 2: number analyzed (Participants) | 1
  Participant 17 Day 2 | 493
  Participant 18 Day 2: number analyzed (Participants) | 1
  Participant 18 Day 2 | 2930

21. Secondary Outcome: Percentage of Participants With Acceptability and Palatability of the Rilematovir Formulation as Assessed by Parent(s)/Caregiver(s)
Description: Acceptability and palatability were assessed by clinician electronic clinical outcome assessment (eCOA) questionnaire which consisted of 7 questions, 1- child took medicine easily, 2- disgusted expressions after tasting medicine, 3- cried after tasting medicine, 4- would not open mouth or turned head away to avoid medicine, 5- spit out or coughed out medicine, 6- gagged, 7- vomited (within 2 minutes of swallowing medicine).
Time Frame: Day 8
Population: ITT-i analysis set included all randomized participants who received at least 1 dose of study intervention and had an RSV infection confirmed by central laboratory analysis. Here, N (Overall number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rilematovir
Number analyzed (Participants) | 7 | 15
Percentage of participants
  Child took medicine easily | 85.7 | 86.7
  Disgusted expressions after tasting medicine | 0 | 13.3
  Did not open mouth or turned head away | 14.3 | 6.7
  Spit out or coughed out medicine | 14.3 | 0
  Gagged | 0 | 6.7
  Vomited (within 2 minutes of swallowing medicine) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Day 35
Description: Safety analysis set included all participants who received at least 1 dose of study intervention.
Arm/Group | Placebo | Rilematovir
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/20
Other Adverse Events (participants affected / at risk) | 5/8 | 10/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | Rilematovir (N=20)
Parainfluenzae Virus Infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | Rilematovir (N=20)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Ventricular Extrasystoles (Cardiac disorders) | 0 (0) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faeces Discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0)
Hyperthermia (General disorders) | 1 (1) | 0 (0)
Infusion Site Extravasation (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Blood Magnesium Decreased (Investigations) | 1 (1) | 0 (0)
Eosinophil Count Increased (Investigations) | 1 (1) | 0 (0)
Oxygen Saturation Decreased (Investigations) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Eczema Infantile (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
As the study was terminated early, the Sponsor decided not to perform the complete analysis planned per protocol. Hence, data was collected and analyzed for safety, and selected PK and efficacy parameters only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/80/NCT04583280/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/80/NCT04583280/SAP_001.pdf